CLINICAL TRIAL: NCT00312169
Title: Evolution of L74V or K65R Mutations in VIremic Subjects on TDF or ABC (EVITA)
Brief Title: Evolution of L74V or K65R Mutations in VIremic Subjects on Tenofovir Disoproxil Fumarate (TDF) or Abacavir (ABC) (EVITA)
Status: Completed | Type: Observational
Sponsor: Orlando Immunology Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Other Study IDs: COL105034 (EVITA); EVITA
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: HIV Infections
Keywords: HIV; NNRTI; Incomplete virologic suppression; treatment experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This is a multicenter, open-label, non-randomized, dual-arm pilot study to investigate the prevalence of the reverse transcriptase (RT) resistance mutations, K65R/x or L74V/x, in HIV-1 plasma from subjects experiencing confirmed first-time incomplete virologic suppression during treatment with an initial antiretroviral (ARV) regimen consisting of at least 12 weeks of TDF or ABC + emtricitabine (FTC) or lamivudine (3TC) + non-nucleoside reverse transcriptase inhibitor (NNRTI) or protease inhibitor (PI). Subjects will be followed until a substantial loss of virologic or immunologic control requires a treatment switch. Confirmed first-time incomplete virologic suppression is defined as an initial plasma HIV-1 RNA response < 400 copies/mL, and subsequent virologic rebound > 400 copies/mL measured at two consecutive times.

Subjects will have a screening genotype to establish adherence to their non-suppressive TDF- or ABC-containing regimen by the presence of M184V (or other treatment-related primary) mutation and to demonstrate that the evolution of treatment-emergent RT mutations can be characterized.

Twenty subjects (a maximum of 10 per arm) will be enrolled at 10-20 United States (U.S.) sites. If fewer than 20 subjects can be enrolled, the study may be discontinued early by the sponsor. Equal numbers of subjects on Arm A versus Arm B will be a goal.

DETAILED DESCRIPTION:
This is a multicenter, open-label, non-randomized, dual-arm pilot study to investigate the prevalence of the RT resistance mutations, K65R/x or L74V/x, in HIV-1 plasma from subjects experiencing confirmed first-time incomplete virologic suppression during treatment with an initial ARV regimen consisting of at least 12 weeks of TDF or ABC + FTC or 3TC + NNRTI or PI. Subjects will be followed until substantial loss of virologic or immunologic control requires a treatment switch. Confirmed first-time incomplete virologic suppression is defined as an initial plasma HIV-1 RNA response < 400 copies/mL, and subsequent virologic rebound > 400 copies/mL measured at two consecutive times.

Subjects will have screening genotype to establish adherence to their non-suppressive TDF- or ABC-containing regimen by the presence of M184V (or other treatment-related primary) mutation and to demonstrate that the evolution of treatment-emergent RT mutations can be characterized.

Twenty subjects (maximum 10 per arm) will be enrolled at 10-20 U.S. sites. If fewer than 20 subjects can be enrolled, the study may be discontinued early by the sponsor. Equal numbers of subjects on Arm A vs. Arm B will be a goal.

Inclusion Criteria

1. Confirmed first-time incomplete virologic suppression during treatment with at least 12 weeks of an ARV regimen consisting of TDF or ABC + FTC or 3TC + NNRTI or PI (TDF as Truvada or individually with FTC, and ABC as Epzicom or individually with 3TC). Confirmed first-time incomplete virologic suppression is defined as an initial plasma HIV-1 RNA response < 400 copies/mL, and subsequent virologic rebound > 400 copies/mL measured at two consecutive times.
2. Screening HIV-1 RNA < 20,000 copies/mL obtained within 30 days prior to study entry.
3. Screening CD4 cell count ≥ 200 cells/mL.
4. Screening HIV-1 genotype with M184V or at least one treatment-related primary mutation.
5. Routine labs as demonstrated by last available lab panel to be:

   * Hemoglobin > 8.0 g/dL;
   * Platelet count > 50,000/mm3;
   * AST (SGOT) < 210 U/L;
   * ALT (SGPT) < 240 U/L;
   * Alkaline phosphatase < 625 U/L;
   * Total bilirubin < 3.25 mg/dL; and
   * Calculated creatinine clearance ≥ 50 as estimated by the Cockcroft-Gault equation.
6. If participating in sexual activity that could lead to pregnancy, female study subjects must use two forms of contraception, one of which must be a barrier method.
7. Men and women aged ≥ 18 years.
8. Ability and willingness of subjects to give written informed consent.

Exclusion Criteria

1. Subjects with screening HIV-1 genotype that is wild-type or contains the resistance mutations K65R/x or L74V/x.
2. Prior or current treatment with ARV regimen consisting of only nucleoside reverse transcriptase inhibitors (NRTIs), zidovudine (ZDV) or stavudine (d4T), more than 2 NRTIs, ritonavir-boosted or dual PI regimen.
3. Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry. Chronic treatment with prednisone at a daily dose of 10 mg or less is permitted. For non-serious illnesses, treatment of less than 21 days with larger doses of corticosteroids is permitted.
4. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
5. Serious illness requiring systemic treatment and/or hospitalization until subject either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 7 days prior to study entry. NOTE: Oral candidiasis, vaginal candidiasis, mucocutaneous herpes simplex, and other minor illnesses (as judged by the site investigator) have no restrictions.
6. Unable to discontinue contraindicated current medications.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed first-time incomplete virologic suppression during treatment with at least 12 weeks of an ARV regimen consisting of TDF or ABC + FTC or 3TC + NNRTI or PI (TDF as Truvada or individually with FTC, and ABC as Epzicom or individually with 3TC). Confirmed first-time incomplete virologic suppression is defined as an initial plasma HIV-1 RNA response < 400 copies/mL, and subsequent virologic rebound > 400 copies/mL measured at two consecutive times.
2. Screening HIV-1 RNA < 20,000 copies/mL obtained within 30 days prior to study entry.
3. Screening CD4 cell count ≥ 200 cells/mL.
4. Screening HIV-1 genotype with M184V or at least one treatment-related primary mutation.
5. Routine labs as demonstrated by last available lab panel to be:

   * Hemoglobin > 8.0 g/dL;
   * Platelet count > 50,000/mm3;
   * AST (SGOT) < 210 U/L;
   * ALT (SGPT) < 240 U/L;
   * Alkaline phosphatase < 625 U/L;
   * Total bilirubin < 3.25 mg/dL; and
   * Calculated creatinine clearance ≥ 50 as estimated by the Cockcroft-Gault equation.
6. If participating in sexual activity that could lead to pregnancy, female study subjects must use two forms of contraception, one of which must be a barrier method.
7. Men and women aged ≥ 18 years.
8. Ability and willingness of subjects to give written informed consent.

Exclusion Criteria:

1. Subjects with screening HIV-1 genotype that is wild-type or contains the resistance mutations K65R/x or L74V/x.
2. Prior or current treatment with ARV regimen consisting of only NRTIs, ZDV or d4T, more than 2 NRTIs, ritonavir-boosted or dual PI regimen.
3. Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry. Chronic treatment with prednisone at a daily dose of 10 mg or less is permitted. For non-serious illnesses, treatment of less than 21 days with larger doses of corticosteroids is permitted.
4. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
5. Serious illness requiring systemic treatment and/or hospitalization until subject either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 7 days prior to study entry. NOTE: Oral candidiasis, vaginal candidiasis, mucocutaneous herpes simplex, and other minor illnesses (as judged by the site investigator) have no restrictions.
6. Unable to discontinue contraindicated current medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin DeJesus, MD, FACP, Study Director — OIC
Locations (11):
- United States (11):
  - Special Services Adult HIV Clinic, Fresno, California
  - AltaMed Health Services Corporation, Los Angelos, California
  - Shared Medical Research Foundation, Tarzana, California
  - Tarzana Treatment Center, Tarzana, California
  - Orlando Immunology Center, Orlando, Florida
  - Northstar Medical Center, Chicago, Illinois
  - Paul Benson, DO, PC, Berkley, Michigan
  - Ricky Hsu, MD, New York, New York
  - Temple University School of Medicine, Section of Infectious Diseases, Philadelphia, Pennsylvania
  - Greenville Hospital System Infectious Disease Associates, Greenville, South Carolina
  - Nicholas C. Bellos, MD PA and Associates, Dallas, Texas